CLINICAL TRIAL: NCT06029530
Title: Delaying the Onset of Nearsightedness Until Treatment Study
Acronym: DONUT
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: sIRB determined feasibility study could not be done because of no benefits of the treatment drops in short time violated FDA requirements
Sponsor: Ohio State University (Other)
Collaborators: University of Houston (Other); State University of New York (Other); Pennsylvania College of Optometry (Industry); Southern California College of Optometry at Marshall B. Ketchum University (Other); University of California, Berkeley (Other); Stanford University (Other); Case Western Reserve University (Other); Illinois College of Optometry (Other); Indiana University (Other); New England College of Optometry (Other); University of the Incarnate Word (Other); Southern College of Optometry (Other); University of Missouri, St. Louis (Other)
Responsible Party: Principal Investigator, Jeffrey J. Walline, OD PhD, Associate Dean for Research, College of Optometry, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: DONUT
Record Dates: First submitted 2023-08-24; First posted 2023-09-08 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Intervention Model Description: Participants will receive one of three concentrations of atropine (0.01%, 0.03%, or 0.05%)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: De-identified bottles will be sent to the sites with randomization codes. The key will be kept at the data coordinating center.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- 0.01% Atropine (Active Comparator): 0.01% atropine eye drops
  Interventions: Drug: Atropine Ophthalmic
- 0.03% Atropine (Active Comparator): 0.03% atropine eye drops
  Interventions: Drug: Atropine Ophthalmic
- 0.05% atropine (Active Comparator): 0.05% atropine eye drops
  Interventions: Drug: Atropine Ophthalmic

INTERVENTIONS:
Drug: Atropine Ophthalmic — eye drops to be administered once daily

SUMMARY:
Participants eligible for the study will be randomized to one of three concentrations of atropine and followed for a month.

DETAILED DESCRIPTION:
Participants will be identified through screening that fit the criteria of a pre-myopic child, which will depend on age and the amount of refractive error at that time. These children will be randomized for a pilot study measuring compliance in nightly eye drop administration. The outcome will be thirty days after randomization, and will assess whether or not there is a difference in compliance between one of three dosages of atropine (0.01%, 0.03%, and 0.05%).

ELIGIBILITY:
Inclusion Criteria:

* Age: 6-11 years
* Refractive error measured in spherical equivalent, one eye meets criterion

  * 6 years old: 0.50 to +0.38
  * 7 years old: 0.50 to +0.25
  * 8-11 years old: 0.50 to plano
* Anisometropia: spherical equivalent <1.50 D
* Astigmatism: <1.50 in both eyes
* Myopia: Less myopic than -0.74 D, both eyes

Exclusion Criteria:

● Myopic

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Compliance percentage | 30 days
  A comparison of the compliance percentage with eye drop administration

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey J Walline, OD PhD, Study Chair — Ohio State University

IPD SHARING:
Plan to Share IPD: No